CLINICAL TRIAL: NCT06501196
Title: A Phase 1/1b Open-Label, Dose Escalation, First-in- Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Anti-leukemic Activity of the Orally Available CDC-Like Kinase (CLK) Inhibitor, BH-30236, in Adults With Relapsed or Refractory Acute Myelogenous Leukemia (R/R AML) or Higher-Risk Myelodysplastic Syndrome (HR-MDS)
Brief Title: A Study of BH-30236 in Relapsed/ Refractory Acute Myelogenous Leukemia and Higher Risk Myelodysplastic Syndrome
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BlossomHill Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BH-30236-01
Record Dates: First submitted 2024-06-17; First posted 2024-07-15 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Leukemia; Leukemia, Myeloid; Leukemia, Myeloid, Acute; Preleukemia; Myelodysplastic Syndromes; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid; Leukemia, Myeloid, Acute; Preleukemia; Myelodysplastic Syndromes | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation Cohort - Monotherapy (Experimental): BH-30236 Monotherapy for Dose Escalation
  Interventions: Drug: BH-30236
- Dose Escalation Cohort - Combination with Venetoclax (Experimental): BH-30236 in Combination with Venetoclax for Dose Escalation.
  Interventions: Drug: BH-30236; Drug: Venetoclax
- Dose Expansion Cohort - Monotherapy (Experimental): BH-30236 based on Monotherapy dose escalation data.
  Interventions: Drug: BH-30236
- Dose Expansion Cohort - Combination with Venetoclax (Experimental): BH-30236 in Combination with Venetoclax based on Dose Escalation data
  Interventions: Drug: BH-30236; Drug: Venetoclax

INTERVENTIONS:
Drug: BH-30236 — BH-30236 will be provided as either a 5 mg, 15 mg or 30 mg tablet. Participants will take BH-30236 tablets orally depending on their dose level assignment.
Drug: Venetoclax — Venetoclax will be provided as 10 mg, 50 mg or 100 mg tablets. Participants will take venetoclax orally per label instructions.
  Other Names: venclexta, venclyxto
  Arms: Dose Escalation Cohort - Combination with Venetoclax; Dose Expansion Cohort - Combination with Venetoclax

SUMMARY:
Study BH-30236-01 is a first-in-human (FIH), Phase 1/1b, open-label, dose escalation and expansion study in participants with relapsed/refractory acute myelogenous leukemia (R/R AML) or higher-risk myelodysplastic syndrome (HR-MDS).

Phase 1, Part 1 Dose Escalation - Monotherapy will evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary efficacy of BH-30236 administered orally. Approximately 50 participants may be enrolled in Phase 1, Part 1 Dose Escalation - Monotherapy.

Phase 1, Part 2 Dose Escalation - Combination with Venetoclax will evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary efficacy of BH-30236 administered as a combination therapy with venetoclax. Approximately 48 participants may be enrolled in Phase 1, Part 2 Dose Escalation - Combination with Venetoclax.

Phase 1b (Dose Expansion) will follow Phase 1 to further understand the relationships among dose, exposure, toxicity, tolerability, and clinical activity. Up to 72 participants may be enrolled in Phase 1b of the study as a monotherapy or in combination with venetoclax.

DETAILED DESCRIPTION:
This is a Phase 1/1b, multi-center, open-label, dose escalation, first-in-human study to evaluate the safety, tolerability, PK, PD, and preliminary anti-leukemic activity of the CLK inhibitor, BH-30236 as a monotherapy or in combination with venetoclax, in adult participants with R/R AML or HR-MDS.

The study consists of three parts: Phase 1, Part 1 Dose Escalation - Monotherapy, Phase 1, Part 2 Dose Escalation - Combination with Venetoclax, and Phase 1b Dose Expansion.

Phase 1, Part 1 Dose Escalation - Monotherapy is anticipated to enroll approximately 50 participants to evaluate the safety, tolerability, PK, PD, and preliminary anti-leukemic activity of BH-30236, as well as determine the MTD and/or the preliminary recommended dose(s) for expansion (RDEs).

Phase 1, Part 2 Dose Escalation - Combination with Venetoclax is anticipated to enroll approximately 48 participants to evaluate the safety, tolerability, PK, PD, and preliminary anti-leukemic activity of BH-30236, as well as determine the MTD and/or the preliminary recommended dose(s) for expansion (RDEs).

Phase 1 will follow a Bayesian optimal interval (BOIN) design dose escalation, where participants will receive ascending doses of BH-30236 to determine the recommended RDEs.

Phase 1b Dose Expansion will enroll approximately 72 participants to evaluate the safety, tolerability, and preliminary anti-leukemic activity of BH-30236 as a monotherapy or in combination with venetoclax at selected RDEs determined in Phase 1 Dose Escalation.

ELIGIBILITY:
Inclusion criteria:

* ≥18 years.
* Diagnosis of relapsed/refractory acute myelogenous leukemia (R/R) AML or higher-risk myelodysplastic syndrome (HR-MDS) with ≥5% bone marrow blast at time of inclusion.
* Prior treatment history must include 1-5 prior lines of therapy.
* ECOG performance status ≤2.
* Adequate organ function evidenced by the following laboratory values:
* Hepatic: Transaminase levels aspartate aminotransferase [AST]/ alanine transaminase [ALT] ≤ 2.5 × upper limit of normal (ULN). In cases of liver involvement by AML or MDS, AST and ALT < 5.0 × ULN is acceptable. Total bilirubin ≤ 1.5 × ULN in the absence of documented Gilbert's disease.
* Renal: Measured or calculated creatinine clearance ≥ 60 mL/min (Cockcroft-Gault formula)

The above are a summary, other inclusion criteria details may apply.

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia or chronic myeloid leukemia with blast crisis.
* Prior allogeneic HSCT within 3 months or donor lymphocyte infusion within 30 days of start of therapy;
* Active and uncontrolled infections.
* Unresolved AEs greater than Grade from prior therapies.
* History of other active malignancy (with certain exceptions)
* Prior treatment with a CLK inhibitor.
* Any acute or chronic graft versus host disease requiring systemic therapy within 4 weeks prior to study drug administration with the exception of topical steroids or the equivalent of 20 mg of prednisone or less.

The above is a summary, other exclusion criteria details may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation: Frequency of dose limiting toxicities (DLTs) | Dose-limiting toxicities are collected during the first treatment cycle (28 days)
  DLTs are dose-limiting toxicities as defined in the study protocol.
Dose Escalation and Expansion: Safety evaluation of BH-30236: Number of participants with treatment-related adverse events as assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | From first dose until 28 days after last dose of BH-30236
  Frequency, severity and relationship to study drug of AEs and SAEs
Dose Expansion: Composite Complete Remission (CR) Rate | From first dose of BH-30236 until disease progression (up to approximately 1 year)
  Composite CR rate disease assessment in accordance with the following guidelines: European Leukemia Network (ELN) 2022 for acute myelogenous leukemia (AML) and International Working Group (IWG) 2023 for myelodysplastic syndrome (MDS).

SECONDARY OUTCOMES:
Dose Escalation and Expansion: Maximum observed blood concentration (Cmax) of BH-30236. | Evaluation performed in Cycle 1 (cycle duration is 28 days).
  Blood samples for PK analyses will be collected at predetermined time points and analyzed.
Dose Escalation: Area under the blood concentration time curve (AUC) of BH-30236. | Evaluation performed in Cycle 1 (cycle duration is 28 days).
  Blood samples for PK analyses will be collected at predetermined time points and analyzed.
Dose Escalation and Expansion: Concentration before dose at steady state (Ctrough). | Evaluation performed in all treatment cycles up to one year (cycle duration is 28 days).
  Blood samples for PK analyses will be collected at predetermined time points and analyzed.
Dose Escalation and Expansion: Objective Response Rate (ORR) | From first dose of BH-30236 until disease progression (up to approximately 1 year)
  Objective response rate disease assessments in accordance with the following guidelines: ELN 2022 recommendations for AML and IWG 2023 for MDS (CR, CR with partial hematologic recovery [CRh], CR with incomplete count recovery [CRi], CR with limited count recovery [CRL], morphologic leukemia-free state [MLFS], or partial response [PR]).
Dose Escalation and Expansion: Duration of Response (DoR) | Time from first documented response until disease progression or death (approximately 1 year).
  Time from first documented response until the date of relapse or death.
Dose Escalation and Expansion: Time to remission (TTR) | From first dose of BH-30236 until complete remission, disease progression or death (approximately 1 year).
  Time from first dose to the achievement of first remission Disease assessments will follow the following guidelines: ELN 2022 for AML and IWG 2023 for MDS.
Dose Escalation and Expansion: Relapse-free Survival (RFS) | From first dose of BH-30236 until disease progression, death, or initiation of a new anti-leukemic therapy (approximately 1 year).
  The time from the start of treatment date to disease progression, death, or initiation of a new anti-leukemic therapy.
Dose Escalation and Expansion: Measurable Residual Disease (MRD) | From time of first dose until discontinuation of BH-30236 (approximately 1 year).
  For AML, using ELN 2022 criteria for disease assessment from Screening, then at the beginning of Cycle 2 and 3, and then every second cycle thereafter.
Dose Escalation and Expansion: Measurement of the change in RNA alternative splicing markers on BH-30236 treatment | From time of first dose until discontinuation of BH-30236 (approximately 1 year).
  Peripheral blood samples for pharmacodynamic (PD) analyses will be collected at predetermined time points and analyzed.
Dose Escalation and Expansion: Complete remission (CR) / complete remission with partial hematologic recovery (CRh) rate for AML and complete remission/partial remission (CR/PR) rate for HR-MDS | Time from first documented response until disease progression or death (approximately 1 year)
  In accordance with the following guidelines: ELN 2022 recommendations for AML and IWG 2023 for MDS (CR, CR with partial hematologic recovery [CRh], CR with incomplete count recovery [CRi], CR with limited count recovery CRL, morphologic leukemia-free state [MLFS], or partial response [PR])

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor Contact, Study Director — BlossomHill Therapeutics, Inc.
Locations (13):
- United States (13):
  - City of Hope Medical Center, Duarte, California
  - University of California Los Angeles, Los Angeles, California
  - Stanford Cancer Center, Palo Alto, California
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern Medicine - Northwestern Memorial Hospital Galter Pavilion, Chicago, Illinois
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Ohio State University Wexner Medical Center - James Cancer Hosp, Columbus, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No